CLINICAL TRIAL: NCT03342365
Title: Evaluation of Intestinal Bacterial and Fungal Translocation and Intestinal Microbiota in Febrile Neutropenic Patients in Pediatric Onco-hematology
Acronym: TRANSNEUTROFEB
Status: Terminated | Type: Observational
Why Stopped: 10 patients inclued instead of 50
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2017/JPL-01
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia | interventions — Microbiota

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Evaluation of microbial translocation and microbiota — Blood test from catheter already in place to determine microbial translocation and stool sample taken for microbiota analysis

SUMMARY:
This pilot study aims to study intestinal bacterial and fungal translocation and the evolution of the intestinal microbiota in patients over the course of their medical surveillance to search for a link between dysbiosis and bacterial/fungal translocation, but also to better understand the elements involved in febrile episodes in these patients (lack of detection of blood microorganisms, translocation of constituent elements of these microorganisms, etc.). We hypothesize that the composition of the intestinal microbiota as well as the phenomenon of intestinal microbial translocation will have an influence on the occurrence of fever and/or bacteremia in neutropenic patients hospitalized in pediatric onco-hematology.

ELIGIBILITY:
* Inclusion Criteria:

  * Information concerning the study set-up, objectives, constraints and the patient's rights is transmitted
  * The patient and/or their legal guardian must have given their free and informed consent. If the patient is over 18, it is the patient who signs the consent form
  * The patient must be a member or beneficiary of a health insurance plan
* Exclusion Criteria:

  * The patient is under state guardianship or safeguard of justice
  * Refusal to sign the consent
  * It is impossible to give the subject informed information
  * Pregnant, parturient or breast feeding patient

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presenting to the CHU Nîmes onco-pediatric service with febrile neutropenia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of presence of bacterial and fungal translocation on occurrence of episodes of febrile neutropenia in pediatric onco-hematology patients. | Between day 7-15
  Presence or absence of microbial translocation; presence = ≥ 10 copies of rDNA16S/µL and/or ≥ 1 copies rDNA 18S/µL and ≥10 ng/mL LBP, ≥10 ng/mL of sCD14 and ≥5 ng/mL of zonulin.

SECONDARY OUTCOMES:
Evaluate prognostic quality of fungal and bacterial translocation markers in occurrence of episodes of febrile neutropenia of unknown origin | Between day 7-15
Evaluate prognostic quality of fungal and bacterial translocation markers in occurrence of episodes of febrile neutropenia in bacteremic patients | Between day 7-15
Compare bacterial and fungal translocation kinetics in febrile neutropenic patients of unknown origin versus bacteremic patients | Between day 7-15
Compare direct (16S rDNA, 18S rDNA) versus indirect (LBP, sCD14 and plasma zonulin) measures of translocation and association with bioclinical characteristics of the population | Between day 7-15
Describe the kinetics of markers and intestinal microbial phylogenetic compositions according to the bioclinical characteristics of the population | Between day 7-15
  Diversity defined by number of different species and number of different taxonomic groups
Creation of biobank | end of study day 30
  All blood and stool samples taken from patients who develop neutropenia. Patients who do not develop neutropenia will have their samples collected at inclusion destroyed

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lavigne, Principal Investigator — CHU Nimes
Locations (3):
- France (3):
  - UFR de Pharmacie Laboratoire de Parasitologie et Mycologie Médicale, Montpellier
  - CHU de Montpellier, Montpellier
  - CHU Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No